CLINICAL TRIAL: NCT02185495
Title: Screening and Diagnosing for Early Lung Cancer in Shanghai Communities With Imaging Procedures
Brief Title: Screening for Early Lung Cancer in Shanghai, China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Fudan University (Other); Ruijin Hospital (Other); Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Principal Investigator, Liu ShiYuan, Shanghai Changzheng Hospital, Shanghai Changzheng Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 13411950100
Record Dates: First submitted 2014-07-05; First posted 2014-07-09 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-11

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-risk individuals (Experimental): The elder and heavy smokers, which are high-risk individuals for early lung cancer. These subjects will be examined using "Observer nodule detection" and " Computer-aided nodule detection".
  Interventions: Behavioral: Observer nodule detection; Device: Computer-aided nodule detection

INTERVENTIONS:
Behavioral: Observer nodule detection — Radiologists will detect the nodules.
Device: Computer-aided nodule detection — Computed-aided detection (CAD) software will be used to detect the nodules.

SUMMARY:
Imaging procedures including chest X-ray and low-dose computed tomography may be effective in lung cancer early detection. Yet it is unknown whether low-dose computed tomography combined with computer aided detection （CAD) is more effective than LDCT in screening of early lung cancer.

DETAILED DESCRIPTION:
The randomized clinical trial is to investigate and compare the effectiveness of CAD-guided low-dose computed tomography and low-dose computed tomography in lung cancer screening for community individuals in Shanghai, China. Thus, an imaging protocol which can detect early lung cancer in asymptomatic high risk patients will be proposed.

ELIGIBILITY:
Inclusion Criteria:

* Age of 55 to 74 years; smoking history of at least 30 pack-years; and if former smoker, have quit within 15 years
* Age 50 or older ,20 or more pack-year history of smoking, and one additional risk factor (occupational exposure, residential radon exposure, cancer history, family history of lung cancer, history of lung disease)
* Age 35 and one additional risk factor
* Ability to accept LDCT examination and sign informed consent form

Exclusion Criteria:

* Individuals with any symptoms suggestive of lung cancer （e.g., vigorous coughing, chest pain, weight loss, blood-stained sputum）
* Individuals with acute pulmonary abnormalities or those in poor health conditions or those have metallic implants or devices in the chest or back will be excluded due to the potential impact on the results as well as difficulty of acquiring the images.
* Pregnant women

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-09 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
The sensitivities of low-dose computed tomography and low-dose computed tomography with computer aided detection in detecting early lung cancer | 24months
  A questionaire will be recorded for each subject, including demographics, smoking history and disease history, etc. If a pulmonary nodule was found, the location, shape, size, margin and density will be recorded.
  A subject with a suspected malignant nodule, which was detected either by a radiologist or computed-aiding detection software, will refer to a physician for further management.
  Finally, the sensitivities of radiologist or software detection will be calculated.

SECONDARY OUTCOMES:
The false positive rates between low-dose computed tomography and low-dose computed tomography with computer aided detection will be compared | 24months
Nodule detection rate | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Shiyuan Liu, MD, Study Director — Radiology Department of Shanghai Changzheng Hospital
Locations (1):
- Changzheng Hospital, Shanghai, Shanghai Municipality, China